CLINICAL TRIAL: NCT03873909
Title: Bioavailability of Carotenoids Present in Mamey Sapote (Pouteria Sapota (Jacq.) H. E. Moore & Stearn) Fruit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hohenheim (Other)
Collaborators: Universidad de Costa Rica (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Sapote2017
Record Dates: First submitted 2019-02-25; First posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Biological Availability
Keywords: Ketocarotenoids; Mamey sapote; Sapotexanthin; Cryptocapsin; Vitamin A

STUDY DESIGN:
Intervention Model Description: randomized 2-way cross-over
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fruit Smoothie (Active Comparator): Post-prandial study feeding 155-200 g mamey sapote mesocarp, 6 g of soybean oil , crushed ice and 150-200 g of water to reach a total volume of 450 mL. (845 µg sapotexanthin, 1.21-1.51 mg cryptocapsin).
  Interventions: Other: Fruit Smoothie
- Matrix-Free Shake (Active Comparator): Post-prandial study feeding 2 g of carotenoid powder formula (845 µg sapotexanthin, 1.21-1.51 mg cryptocapsin), 37.5 g of sugar, 75 µg of citric acid, 6 g of soybean oil emulsified into 300 g of water using 3 g of soy lecithin as well as ca. 100 g of crushed ice, yielding a shake volume of 450 mL.
  Interventions: Other: Matrix-Free Shake

INTERVENTIONS:
Other: Fruit Smoothie — Fruit Smoothie with 150-200 g mamey sapote fruit
  Arms: Fruit Smoothie
Other: Matrix-Free Shake — Shake containing mamey sapote extracted carotenoids (2 g, 845 µg sapotexanthin and 1.21-1.51 mg cryptocapsin
  Arms: Matrix-Free Shake

SUMMARY:
The goal of the study is to determine if mamey sapote fruit, rich in rare potentially provitamin A keto-carotenoids, is a good source of vitamin A in humans. Furthermore, it will help to compare the absorption of carotenoids between the fruit versus a "matrix-free" formulation.

The objective will be accomplished by quantitation of the immediate post-prandial plasma concentrations of parent carotenoids and vitamin A metabolites from participants consuming a meal consisting of a mamey sapote fruit smoothie or a shake containing mamey sapote encapsulated carotenoids.

DETAILED DESCRIPTION:
The present study seeks to obtain a better understanding of the bioavailability and metabolism of the exceptional keto-carotenoids, sapotexanthin and cryptocapsin from mamey sapote fruit in humans. For this purpose, the absorption of such carotenoids after the consumption of fresh mamey sapote fruit and a "matrix-free" water-dispersible formulation containing isolated mamey sapote carotenoids will be compared.

The participants of the study will be healthy, non-pregnant, non-smoking adults aged 18-65. Prior to the study, the people who wants to participate in the study will have an education session where the coordinator explains the study in detail and discusses which foods and supplements need to be avoided during the study. They will give their consent to participate in the study, will be screened for body height/weight (BMI) and will complete a health questionnaire. Afterward, if they fit the necessary health criteria for the study, they will be enrolled as a participant and an appointment will be made for their post-prandial visit to the School of Medicine (University of Costa Rica).

The participants will refrain from consuming products containing high levels of carotenoids (β-carotene, β-cryptoxanthin, lutein, and zeaxanthin) for 10 days prior to the first day of treatment until the end of the study ("washout"). They will receive a list of foods and supplements to avoid. They will record their actual daily consumption of carotenoid-containing foods on the list of foods to avoid. The record will allow determining whether participants are remaining compliant and avoiding carotenoid-containing foods.

For the post-prandial visit, a blood sample will be taken at hour 0 (baseline sample) and then the corresponding test meal (fruit smoothie or matrix-free shake) will be administered to the participants. Subsequent blood sampling will be carried out at 2,4,5,6,8 and 9.5 h after the meal is consumed. A carotenoid-free lunch will be provided at 4.5 hours. Afterward, the triglyceride-rich fraction (TRL) will be isolated from the plasma samples and the concentration of carotenoids and retinyl esters determined. The values obtained will be used to determine the mean value of the Area Under the Curve (AUC) through time to compare the absorption between the two meals provided.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult men and women with a BMI 17 to 30
* Aged 18-65 years.

Exclusion Criteria:

* lactating, pregnant, or planned to be pregnant
* smokers/those who use tobacco products
* metabolic or malabsorption disorders
* with history of cancer
* with history of liver insufficiency or other gastro-intestinal diseases
* with history of chronic diseases related to lipid metabolism
* obesity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2017-11-13 (Actual); Study Completion 2018-03-13 (Actual)

PRIMARY OUTCOMES:
Change in carotenoid concentration in blood plasma over 9.5 h after meal consumption | 7 post-prandial blood samples over 9.5 hours including baseline
  An area under the curve for concentration of carotenoids (from triglyceride-rich lipoprotein (TRL) fraction of plasma) will be obtained by using carotenoid concentrations from hours 0, 2, 4, 5, 6, 8 and 9.5 over time to quantify absorption after subjects consume a meal consisting of a mamey sapote fruit smoothie or a "matrix-free" carotenoid-rich shake.
Change in retinyl esters concentration in blood plasma over 9.5 h after meal consumption | 7 post-prandial blood samples over 9.5 hours including baseline
  An area under the curve for concentration of retinyl esters (from triglyceride-rich lipoprotein (TRL) fraction of plasma) will be obtained by using retinyl esters concentrations from hours 0, 2, 4, 5, 6, 8 and 9.5 over time to quantify conversion of carotenoids to retinyl esters after subjects consume a meal consisting of a mamey sapote fruit smoothie or a "matrix-free" carotenoid-rich shake.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Esquivel, Ph.D, Principal Investigator — Universidad de Costa Rica; Silvia Quesada, Principal Investigator — Universidad de Costa Rica
Locations (2):
- University of Costa Rica, San José, San Pedro de Montes de Oca, Costa Rica
- University of Hohenheim, Stuttgart, Germany

IPD SHARING:
Plan to Share IPD: No